CLINICAL TRIAL: NCT02715622
Title: A Prospective, Multicenter Post-Market Study to Evaluate and Compare the Clinical Outcomes, Pain and Patient Quality of Life After Open, Laparoscopic or Robotic Assisted Hernia (Incisional and Inguinal) Repair
Brief Title: A Prospective Study to Compare the Clinical Outcomes, Pain and Patient Quality of Life for Hernia Patients
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Collaborators: Accelovance (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-PHS-2016
Record Dates: First submitted 2016-02-19; First posted 2016-03-22 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hernia; Incisional Hernia; Hernia, Inguinal, Indirect; Hernia, Inguinal, Direct; Inguinal Hernia
MeSH Terms: conditions — Hernia; Incisional Hernia; Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Open Hernia Repair: A minimum of 300 patients will be enrolled in the Incisional and Inguinal Hernia open repair surgical procedure
  Interventions: Procedure: Hernia repair
- Laparoscopic Hernia Repair: A minimum of 300 patients will be enrolled in the Incisional and Inguinal Hernia laparoscopic repair surgical procedure
  Interventions: Procedure: Hernia repair
- Robotic Hernia Repair: A minimum of 300 patients will be enrolled in the Incisional and Inguinal Hernia robotic-assisted laparoscopic repair surgical procedure
  Interventions: Procedure: Hernia repair

INTERVENTIONS:
Procedure: Hernia repair — Patient undergoing Hernia repair using different surgical modalities as per the surgeon's standard of care practice

SUMMARY:
The objective of this prospective, multi-center post-market study is to prospectively collect uniform, evidence based outcomes for patients undergoing open, laparoscopic or robotic assisted hernia repair.

The outcomes that will be collected include various routine clinical parameters, short term patient reported outcomes (quality of life, pain scores) and long term hernia recurrence information. Patients will be treated according to standard of care at the surgeon's institution and patients will be followed up to collect information related to complications information and patient satisfaction associated with the hernia repair procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. All patients undergoing either an open, laparoscopic or robotic-assisted
3. Incisional or Inguinal Hernia repair procedure
4. Non-Emergent Incisional or Inguinal Hernia Repair cases

Exclusion Criteria:

1. Emergent Cases for both Incisional and Inguinal Hernia
2. Incisional Hernia related to ostomy formation
3. Incisional Hernia requiring component separation (determined pre-operatively or intraoperatively)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 900 patients will be enrolled in this post-market study that is planned to be conducted for mainly 2 types of hernia repairs, Incisional hernia repair and inguinal hernia repair ( robotic-assisted, lap and open). Up to 2000 patients may be enrolled.
  Approximately 450 patients who will undergo inguinal hernia repair across open, laparoscopic or robotic-assisted procedures (~ 150 patients in each surgical modality) and approximately 450 patients who will undergo incisional hernia repair across open, laparoscopic or robotic-assisted procedures (~ 150 patients in each surgical modality) will be enrolled in this study at up to thirty (30) study centers
Sampling Method: Non-Probability Sample
Enrollment: 944 (Actual)
Dates: Start 2016-04; Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Number of complications observed intraoperatively through 30 days | 30 days
  Number of intraoperative and short-term complications related to hernia repair.
Number of patient reported complications post 30-days through 3 years post procedure | 30 days post-procedure to 3 years post-procedure
  Number of long-term complications related to hernia repair directly reported by patients

SECONDARY OUTCOMES:
Patient reported outcomes on Quality of Life through 1 year | Pre-procedure (baseline) and 30 days through 1 year for Qualify of Life
  Use of quality of life questionnaires (Carolinas Comfort Scale or HerQles Abdominal Questionnaire) will be used to assess patient qualify of life pre-procedure and post-procedure through 1 year.
Incisional or Inguinal Hernia Recurrence through 3 years | 30 days post-procedure through 3 years
  Number of hernia recurrences for each patient will be patient reported through 3 years post-procedure.
Patient reported outcomes on post-procedure pain through 3 years | 2-4 weeks post-procedure through 3 years post-procedure
  Pain medication taken by patient (type, dosage and quantity of pills) will also be captured through patient reported methods. Unit of measure will be numerical count of pills take

CONTACTS AND LOCATIONS:
Overall Officials: Karl LeBlanc, MD, Study Chair — Surgeon Group of Baton Rouge
Locations (17):
- United States (17):
  - Beverly Hills Hernia Center, Beverly Hills, California
  - Vanderbilt University Medical Center, Nashville, California
  - Kaiser Foundation Research Institute, Oakland, California
  - Florida Hospital - Celebration Health, Celebration, Florida
  - Baptist Health South Florida, South Miami, Florida
  - Southern Illinois Healthcare, Carbondale, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Progressive Surgical Associates, New Lenox, Illinois
  - Louisville Surgical Associates, Louisville, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Spectrum Health System, Grand Rapids, Michigan
  - The Mount Sinai Medical Center, New York, New York
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - University of Tennessee, Memphis, Tennessee
  - The Dallas VA Research Corporation, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] LeBlanc KA, Gonzalez A, Dickens E, Olsofka J, Ortiz-Ortiz C, Verdeja JC, Pierce R; Prospective Hernia Study Group. Robotic-assisted, laparoscopic, and open incisional hernia repair: early outcomes from the Prospective Hernia Study. Hernia. 2021 Aug;25(4):1071-1082. doi: 10.1007/s10029-021-02381-0. Epub 2021 May 24. PMID 34031762
- [Derived] LeBlanc KA. Design of a comparative outcome analysis of open, laparoscopic, or robotic-assisted incisional or inguinal hernia repair utilizing surgeon experience and a novel follow-up model. Contemp Clin Trials. 2019 Nov;86:105853. doi: 10.1016/j.cct.2019.105853. Epub 2019 Oct 25. PMID 31669560